CLINICAL TRIAL: NCT00744419
Title: A Multicenter, Open-label, Single and Multiple Dose Pharmacokinetic Study of IV Pantoprazole in Preterm Infants and Infants 0-11 Months With a Clinical Diagnosis of Gastroesophageal Reflux Disease (GERD) or the Need for Acid Suppression
Brief Title: Intravenous (IV) Pantoprazole for Gastroesophageal Reflux Disease (GERD) in Neonates and Infants
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: University of Louisville (Other)
Collaborators: Wyeth is now a wholly owned subsidiary of Pfizer (Industry)
Responsible Party: Principal Investigator, Janice E. Sullivan, Professor, University of Louisville
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: UofL Panto 01
Record Dates: First submitted 2008-08-29; First posted 2008-09-01 (Estimated); Last update posted 2015-12-03 (Estimated); Status verified 2015-12

CONDITIONS: Gastroesophageal Reflux
Keywords: GERD; pharmacokinetics; pantoprazole; neonates; infants
MeSH Terms: conditions — Gastroesophageal Reflux | interventions — Pantoprazole

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- 3 age groups (Experimental): Assigned to the arm based on age.
  Interventions: Drug: pantoprazole

INTERVENTIONS:
Drug: pantoprazole — Intravenous pantoprazole will be administered daiy for 6 (+/- 1 day). The first 6 subjects in each age group will receive low dose [0.4 mg/kg (< 44 wks PMA) or 0.8 mg/kg (44 wks to < 1 yr)] and the last 6 subjects in each age group will receive high dose [0.8 mg/kg(< 44 wks PMA) or 1.6 mg/kg(44 wks to < 1 yr)]
  Other Names: Protonix

SUMMARY:
The purpose of this study is to determine how the body uses and eliminates pantoprazole, a drug used to treat GERD. This is a pharmacokinetic (PK) study. PK is a measure of how much drug is in the blood and how long it takes to leave the body. It is hypothesized that younger infants will need a lower dose than older children to achieve the same PK measurement.

The results of this study will be used to determine the best dose of the drug to use in each age group. Pantoprazole is a drug used to decrease acid production. The use of pantoprazole has not been approved for use in children. Pantoprazole is approved for use of acid-related and stomach disorders in adults.

DETAILED DESCRIPTION:
Gastroesophageal reflux, regurgitation of gastric contents into the esophagus, and gastroesophageal reflux disease, displaying symptoms and complications from regurgitation, are both very common in infants. Daily reflux is present in up to 50% of infants younger than 3 months and in more than 66% at 4 months of age. GERD is primarily attributed to lower esophageal sphincter relaxation. Between 5-9% of infants less than one year of age have GERD and require acid suppression. Complications associated with GERD include failure to thrive, apnea, wheezing, recurrent aspiration, poor feeding, refusal to feed, irritability, and in more severe cases, acute life-threatening events.

Pantoprazole is a proton pump inhibitor that suppresses the final step in gastric acid production through binding to the H+-K+-ATPase enzyme system at the surface of parietal cells in gastric epithelium. This causes a reduction in acid production regardless of the stimulus presented. Pantoprazole is used as therapy in GERD, erosive esophagitis, gastritis, gastric ulcerations, duodenal ulcerations and prophylaxis of stress gastritis in hospitalized patients. Pantoprazole is metabolized mainly by hepatic cytochrome P-450 CYP2C19 and is hypothesized to be metabolized at a higher rate in children as compared to adults. However, the metabolism of proton pump inhibitors is slower in infants < 10 weeks of age. Clinical studies are ongoing for the use of oral pantoprazole in infants and children.

Acid suppression is frequently required in hospitalized infants to treat GERD. In children who are critically ill, oral administration of acid suppressive agents is relatively contraindicated therefore an intravenous alternative such as intravenous pantoprazole is imperative. Intravenous pantoprazole has been well tolerated in pharmacokinetic studies in children ages 1 to 16 years. No systematic studies have been done to determine the pharmacokinetics of intravenous pantoprazole in infants less than 1 year of age therefore this study will meet an identified unmet need and address a knowledge deficit in this population. The aim of this study is to determine the pharmacokinetics of pantoprazole sodium for injection and evaluate the safety and tolerability of single and multiple intravenous doses in preterm neonates and infants 0-11 months of age using population pharmacokinetics. In addition, the genotyping for CYP2C19 and CYP3A4 polymorphisms will be performed.

ELIGIBILITY:
Inclusion Criteria:

1. Signed informed consent and HIPAA documents by parent/legal guardian.
2. Hospitalized premature neonates (Post menstrual age (PMA) 28 - < 34 weeks), neonates (PMA 34 to 44 weeks), and infants (PMA > 44 weeks to 11 months).
3. Clinical indication for acid suppression or a presumptive diagnosis of GERD based on clinical symptoms and/or objective tests diagnostic of GERD.
4. Body weight of at least 750 grams (based on blood volume required for study participation).

Exclusion Criteria:

1. Previous adverse reaction to proton pump inhibitor
2. History of gastrointestinal anomalies, eosinophilic esophagitis, unrepaired tracheal esophageal fistula or liver disease
3. Unstable cardiovascular, renal, hepatic, hematologic or endocrine disease
4. History of acute life-threatening events due to GERD
5. History of hepatitis B or hepatitis C
6. Use of PPI's within 24 hours before study drug is administered
7. Known human immunodeficiency virus (HIV) or acquired immune deficiency syndrome
8. Clinically significant laboratory values:

   * Aspartate aminotransferase (AST) or alanine aminotransferase (AST) >2 times the upper limit of normal (ULN) for age
   * Total bilirubin > 2 times ULN for age
   * Alkaline phosphatase > 2 times ULN for age

10.Use of histamine-2 receptor blockers (eg. Cimetidine, famotidine, ranitidine, or nizatidine) sucralfate, misoprostol, or prokinetic agents (eg. urecholine, erythromycin, or metoclopramide) and antacids or bismuth preparations within 24 hours before test article administration.

11.Any disorder requiring chronic use of warfarin, oxcarbazepine, topiramate, carbamezapine, rifampin or phenytoin.

12.Currently participating in another investigational drug trial or have participated in a study within the last 30 days.

Ages: 28 Weeks to 11 Months | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 24 (Actual)
Dates: Start 2009-05; Primary Completion 2012-04 (Actual); Study Completion 2012-04 (Actual)

PRIMARY OUTCOMES:
The primary endpoint is to characterize the pharmacokinetics of intravenous pantoprazole after a single dose and multiple doses in neonates and infants less than one year of age with presumed GERD. | 0, 0.5, 1, 2, 3, 6, 8 and 12 hours (Day 1) and 0, 2, 3 and 4 hours (Day 6) with a maximum of 6 samples per subject. (Each subject will be assigned to a specific PK group)

SECONDARY OUTCOMES:
To describe the safety of pantoprazole in neonates and infants less than one year of age with presumed GERD. To compare the pantoprazole PK data obtained from this study population to data obtained from subjects greater than 1 year of age. | From enrollment to 14 days after the last dose of study drug.

CONTACTS AND LOCATIONS:
Overall Officials: Angela M Jeffries, MD, Principal Investigator — University of Louisville
Locations (1):
- University of Louisville Research Foundation, Inc/KCPCRU, Louisville, Kentucky, United States